CLINICAL TRIAL: NCT00122083
Title: A Cluster Randomised Controlled Trial to Assess the Effectiveness of a Simple Marketing Intervention in Changing Student Attitudes to Depression
Brief Title: An Evaluation of the Effectiveness of a Simple Marketing Intervention in Changing Student Attitudes to Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oxford (Other)
Collaborators: Pfizer (Industry); Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Educational/Counseling/Training
Other Study IDs: UOxford
Record Dates: First submitted 2005-07-18; First posted 2005-07-21 (Estimated); Last update posted 2005-07-26 (Estimated); Status verified 2004-03

CONDITIONS: Depression
Keywords: Depression; Students; Health education
MeSH Terms: conditions — Depression; Health Education

INTERVENTIONS:
Device: Health education information

SUMMARY:
The purpose of this study is to determine the effectiveness of a simple marketing intervention in changing attitudes towards depression and its treatment among university students.

DETAILED DESCRIPTION:
Depression is a major public health problem. It is common, affecting approximately 10 percent of the United Kingdom (UK) community at any one time. Britain's student population is particularly at risk.

Knowledge of effective treatments for depression is burgeoning thanks to a rapid increase in the quantity and quality of relevant research. Regardless of these advances, depression is still under-reported (Freeling et al., 1985) and general practitioners often fail to diagnose it.

When depression is correctly diagnosed, most patients in primary care will receive a prescription for an antidepressant. However, some patients will not have the prescription dispensed, and most will not complete the full recommended course. Compliance with psychological treatments is also a problem.

Study Design:

* Pilot work: The intervention consisted of mailing (to each undergraduate student's pigeon-hole) a pack of 4 postcards which provided brief information on depression in an attractive format. One postcard summarised information on depression as an illness; one summarised information on the causes of depression; one summarised information on the treatment of depression; and one summarised information on how to seek help for depression. Prior to the trial, the drafts were revised through feedback from a focus group of 5 students, who discussed the design and content of the draft postcards. The focus group participants were recruited from the Queen's College, as this college did not participate in the trial. The focus group contributed to the revision of the draft questionnaire.
* The trial: The design was a cluster, randomised, controlled trial. Individual Oxford University colleges which accept undergraduate students were the units of randomisation. Twenty-eight colleges were randomised. Permanent private halls and postgraduate colleges were excluded, as was the Queen's College (due to it being the lead investigator's college) and Harris Manchester College (a college for mature students).

Half of the randomised colleges received no intervention; the other half received the intervention.

A questionnaire was administered before and after the intervention to half of the undergraduate students in each of the colleges. The same questionnaire was used for both time points. Questions addressed knowledge of, and attitudes towards:

* depression as an illness;
* symptoms of depression;
* treatment for depression;
* sources of help for depression.

ELIGIBILITY:
Inclusion Criteria:

* Undergraduate students at Oxford University

Exclusion Criteria:

* Postgraduate students
* Students at the excluded colleges

Min Age: 0 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1680
Dates: Start 2004-04; Study Completion 2004-06

PRIMARY OUTCOMES:
The primary outcome was the proportion of participants responding positively to the question 'Can depression be effectively treated?'

SECONDARY OUTCOMES:
Secondary outcomes included the correct identification of the symptoms of depression and the effectiveness of certain treatments.

CONTACTS AND LOCATIONS:
Overall Officials: John Geddes, Principal Investigator — University of Oxford
Locations (1):
- University of Oxford, Oxford, Oxfordshire, United Kingdom

REFERENCES:
- [Background] Birrer RB. Depression and aging too often do mix. Postgrad Med. 1998 Sep;104(3):143-9, 153-4, 163-4. doi: 10.3810/pgm.1998.09.580. PMID 9742909
- [Background] Freeling P, Rao BM, Paykel ES, Sireling LI, Burton RH. Unrecognised depression in general practice. Br Med J (Clin Res Ed). 1985 Jun 22;290(6485):1880-3. PMID 3924297